CLINICAL TRIAL: NCT01626690
Title: Prospective Randomized Control Trial of the Effect of Preoperative Forced-air Warming on Perioperative Body Temperature Following Neuraxial Anesthesia in Total Hip Arthroplasty Patients
Brief Title: Prospective Trial of the Effect of Preoperative Forced-air Warming on Perioperative Body Temperature Following Neuraxial Anesthesia in Total Hip Arthroplasty Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Surgeons change in preference for perioperative warming.
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0823
Record Dates: First submitted 2012-06-12; First posted 2012-06-25 (Estimated); Results first posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-07

CONDITIONS: Perioperative Hypothermia

ARMS (2):
- Pre-Warming (Experimental)
  Interventions: Device: Bair-Paws Warming Device
- Control (Active Comparator)
  Interventions: Device: Bair-Hugger Warming Device

INTERVENTIONS:
Device: Bair-Paws Warming Device — Bair-Paws device to be applied to patient and used for perioperative (including preoperative) warming.
  Arms: Pre-Warming
Device: Bair-Hugger Warming Device — Bair-Hugger device to be applied to patient and used for intraoperative warming (current standard of care at our institution).
  Arms: Control

SUMMARY:
The purpose of this study is to determine if placement of a forced-air warming device prior to institution of regional anesthesia improves perioperative temperature control in patients undergoing total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing total hip arthroplasty under neuraxial anesthesia,
* age 55-85,
* BMI 18-40

Exclusion Criteria:

* allergy to local anesthetics,
* patients electing to have general anesthesia for their total hip arthroplasty,
* pregnancy,
* prisoners,
* patients unable to give informed consent,
* English as a second language,
* active infectious or febrile illness (measured temperature > 37.5 degrees Celsius).

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pre-Warming | Control
Started | 49 | 51
Completed | 47 | 51
Not Completed | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-Warming | Control | Total
Number analyzed (Participants) | 47 | 51 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 23 | 44
  >=65 years | 26 | 28 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.1 (6.37) | 66.5 (7.41) | 66.3 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 24 | 51
  Male | 20 | 27 | 47
Region of Enrollment [Number; unit: participants]
  United States | 47 | 51 | 98
Baseline Temperature [Mean (Standard Deviation); unit: Degrees Celisius] | 36.6 (0.4) | 36.7 (0.37) | 36.6 (0.39)

OUTCOME MEASURES:

1. Primary Outcome: Patient Temperature at the Time of Incision as Measured by SpotOn (3M) Temperature Monitoring System..
Description: Temporal artery temperature readings (in degrees celsius) will be obtained at the time of incision and every 30 minutes while in the OR.
Time Frame: The treatment period starts with the patient consenting to the study and application of preoperative forced-air warming device and ends when the patient leaves the PACU (average 4-8 hours following enrollment).
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Pre-Warming | Control
Number analyzed (Participants) | 47 | 51
Degrees Celsius | 35.7 (0.47) | 35.4 (0.49)

2. Secondary Outcome: Patient Temperature Prior to Entering OR as Measured by SpotOn (3M) Temperature Monitoring System.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Pre-Warming | Control
Number analyzed (Participants) | 47 | 51
Degrees Celsius | 36.7 (0.4) | 36.6 (0.4)

3. Secondary Outcome: Patient Temperature 30 Minutes Following Incision as Measured by SpotOn (3M) Temperature Monitoring System.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Pre-Warming | Control
Number analyzed (Participants) | 47 | 51
Degrees Celsius | 35.7 (0.4) | 35.4 (0.4)

4. Secondary Outcome: Patient Temperature on Arrival to Recovery Room as Measured by SpotOn (3M) Temperature Monitoring System.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Pre-Warming | Control
Number analyzed (Participants) | 47 | 50
Degrees Celsius | 35.4 (0.8) | 35.1 (0.6)

5. Secondary Outcome: Incidence of Postoperative Shivering in Recovery Room.
Time Frame: as for outcome 1
Measure: Number; unit: Number of patients reporting shivering
Arm/Group | Pre-Warming | Control
Number analyzed (Participants) | 47 | 51
Number of patients reporting shivering | 1 | 14

6. Secondary Outcome: Intraoperative Blood Loss.
Description: Intraoperative blood loss in mL's.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Pre-Warming | Control
Number analyzed (Participants) | 47 | 51
mL | 263 (109) | 307 (116)

7. Secondary Outcome: Incidence of Perioperative Cardiac Events.
Description: Incidence of perioperative arrhythmias or myocardial ischemia.
Time Frame: as for outcome 1
Measure: Number; unit: Patients
Arm/Group | Pre-Warming | Control
Number analyzed (Participants) | 47 | 51
Patients | 1 | 0

8. Secondary Outcome: Temporal Artery Verus SpotOn (3M) Temperature Readings.
Description: Temperature with temporal artery thermometer and SpotOn temperature monitoring device (3M) at time of incision.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Groups:
- Temporal Artery Thermometer: Patient temperature at time of incision as measured by temporal artery thermometer.
- SpotOn (3M) Temperature Readings.: Patient temperature at time of incision as measured by SpotOn (3M) temperature monitoring system.
Arm/Group | Temporal Artery Thermometer | SpotOn (3M) Temperature Readings.
Number analyzed (Participants) | 98 | 98
Degrees Celsius | 36.5 (0.5) | 36.5 (0.5)

ADVERSE EVENTS:
Arm/Group | Pre-Warming | Control
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/51
Other Adverse Events (participants affected / at risk) | 0/47 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes